CLINICAL TRIAL: NCT02857855
Title: The Impact of Postoperative Oxygen Therapy on the Results of Liver Transplantation
Brief Title: Postoperative Supplemental Oxygen in Liver Transplantation
Acronym: PSOLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1WB/1/23/06/2016
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Infection
Keywords: liver transplantation; postoperative infection; biliary complications; patient survival; graft survival; supplemental oxygen
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80% fraction of inspired oxygen (Experimental): 80% fraction of inspired oxygen delivered either by a nonrebreathing facemask with a reservoir with oxygen flow of 14 l/min and air flow of 2 l/min or by a respirator for first 6 postoperative hours
  Interventions: Procedure: 80% fraction of inspired oxygen for 6 postoperative hours
- 28% fraction of inspired oxygen (Active Comparator): 28% fraction of inspired oxygen delivered either by a Venturi facemask or by a respirator for first 6 postoperative hours
  Interventions: Procedure: 28% fraction of inspired oxygen for 6 postoperative hours

INTERVENTIONS:
Procedure: 80% fraction of inspired oxygen for 6 postoperative hours — 80% fraction of inspired oxygen delivered for 6 postoperative hours, either by a nonrebreathing facemask with a reservoir or by a respirator
  Arms: 80% fraction of inspired oxygen
Procedure: 28% fraction of inspired oxygen for 6 postoperative hours — 28% fraction of inspired oxygen delivered for 6 postoperative hours, either by a Venturi facemask or by a respirator
  Arms: 28% fraction of inspired oxygen

SUMMARY:
The aim of this prospective randomized controlled trial is to evaluate the impact of high concentration supplemental postoperative oxygen therapy on short-term and long-term results of liver transplantation, particularly with respect to infections and biliary complications.

DETAILED DESCRIPTION:
The aim of this prospective randomized controlled trial is to evaluate the impact of high concentration supplemental postoperative oxygen therapy on short-term and long-term results of liver transplantation, particularly with respect to infections and biliary complications. A total of 296 patients immediately after liver transplantation will be randomly assigned to receive either 80% (high concentration) or 28% (controls) fraction of inspired oxygen for 6 hours after surgery with a 1:1 allocation ratio. Patients will be blinded to the type of received intervention. Randomization will be stratified by the Child-Turcotte-Pugh classification. Both groups will be compared to short- and long-term outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* active liver transplant waitlist status

Exclusion Criteria:

* active infection at the time of transplantation
* malignancy
* cardiac arrest during transplantation
* chronic obstructive pulmonary disease
* acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative infections | 30 days
  Occurrence of postoperative infection defined according to the Centers for Disease Control and Prevention (Am J Infect Control 2008; 36: 309-32)

SECONDARY OUTCOMES:
Biliary complications | 5 years
  Biliary complications requiring endoscopic, percutaneous or surgical intervention
Postoperative mortality | 90 days
Severe postoperative complications | 90 days
  >= grade 3 according to Clavien-Dindo classification
Patient survival | 5 years
Graft survival | 5 years
Postoperative hospital stay | 1 year
Postoperative intensive care unit stay | 1 year
Serum aspartate aminotransferase activity | 5 days
Serum alanine aminotransferase activity | 5 days
Serum bilirubin concentration | 5 days
International normalized ratio | 5 days
Early allograft dysfunction | 7 days
  One or more of the following: bilirubin >or=10mg/dL on postoperative day 7, international normalized ratio >or=1.6 on postoperative day 7, alanine or aspartate aminotransferases >2000 IU/L within the first postoperative 7 days (Olthoff et al, Liver Transpl 2010; 16: 943-9)
Pulmonary complications | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michał Grąt, M.D., PhD., Principal Investigator — Department of General, Transplant and Liver Surgery, Medical University of Warsaw
Locations (1):
- Department of General, Transplant and Liver Surgery, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the investigators on reasonable request.

REFERENCES:
- [Derived] Figiel W, Niewinski G, Grat M, Krawczyk M, Stypulkowski J, Lewandowski Z, Krasnodebski M, Patkowski W, Zieniewicz K. Postoperative Supplemental Oxygen in Liver Transplantation (PSOLT) does not reduce the rate of infections: results of a randomized controlled trial. BMC Med. 2023 Feb 13;21(1):51. doi: 10.1186/s12916-023-02741-w. PMID 36782227